CLINICAL TRIAL: NCT07350005
Title: A Prospective Randomized Study Comparing the Efficiency and Safety of Holmium:YAG, Thulium:YAG, and Thulium Fiber Lasers in Anatomical Prostate Enucleation
Brief Title: Comparison of Holmium, Thulium:YAG, and Thulium Fiber Lasers in Prostate Enucleation
Acronym: TRI-LASER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, erol maraş, Principal Investigator, Ankara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AUTF-TRI-LASER-01
Record Dates: First submitted 2026-01-06; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: BPH (Benign Prostatic Hyperplasia)
Keywords: bph; prostate; holmium; thulium; TFL
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in parallel to one of three intervention arms corresponding to Holmium:YAG, Thulium:YAG, or Thulium Fiber Laser-based anatomical prostate enucleation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Holmium:YAG Laser Enucleation (Active Comparator): Participants in this arm will undergo anatomical prostate enucleation using Holmium:YAG laser as part of standard surgical treatment for benign prostatic hyperplasia.
  Interventions: Procedure: Holmium:YAG Laser Prostate Enucleation
- Thulium:YAG Laser Enucleation (Active Comparator): Participants in this arm will undergo anatomical prostate enucleation using Thulium:YAG laser as part of standard surgical treatment for benign prostatic hyperplasia.
  Interventions: Procedure: Thulium:YAG Laser Prostate Enucleation
- Thulium Fiber Laser (TFL) Enucleation (Active Comparator): Participants in this arm will undergo anatomical prostate enucleation using Thulium Fiber Laser (TFL) as part of standard surgical treatment for benign prostatic hyperplasia.
  Interventions: Procedure: Thulium Fiber Laser Prostate Enucleation

INTERVENTIONS:
Procedure: Holmium:YAG Laser Prostate Enucleation — Anatomical prostate enucleation performed using a Holmium:YAG laser system as part of standard surgical treatment for benign prostatic hyperplasia.
  Arms: Holmium:YAG Laser Enucleation
Procedure: Thulium:YAG Laser Prostate Enucleation — Anatomical prostate enucleation performed using a Thulium:YAG laser system as part of standard surgical treatment for benign prostatic hyperplasia.
  Arms: Thulium:YAG Laser Enucleation
Procedure: Thulium Fiber Laser Prostate Enucleation — Anatomical prostate enucleation performed using a Thulium Fiber Laser (TFL) system as part of standard surgical treatment for benign prostatic hyperplasia.
  Arms: Thulium Fiber Laser (TFL) Enucleation

SUMMARY:
Benign prostatic hyperplasia (BPH) is a common condition in aging men and may require surgical treatment when medical therapy is ineffective. Anatomical prostate enucleation using different laser technologies is a well-established surgical approach for the treatment of BPH.

The purpose of this prospective randomized study is to compare the efficiency and safety of three commonly used laser systems-Holmium:YAG, Thulium:YAG, and Thulium Fiber Laser (TFL)-during anatomical prostate enucleation.

The primary objective of the study is to evaluate laser efficiency by measuring grams of enucleated prostate tissue per joule (g/J) using intraoperative laser device data. Secondary outcomes include changes in International Prostate Symptom Score (IPSS) and the occurrence of postoperative urinary incontinence.

All laser systems used in this study are part of routine clinical practice, and no additional diagnostic procedures or treatments will be performed for study purposes

DETAILED DESCRIPTION:
This is a prospective, randomized, single-center clinical study designed to compare the efficiency and safety of three different laser systems used in anatomical prostate enucleation for the surgical treatment of benign prostatic hyperplasia (BPH).

Eligible patients will be randomly assigned to undergo prostate enucleation using one of the following laser technologies: Holmium:YAG laser, Thulium:YAG laser, or Thulium Fiber Laser (TFL). All procedures will be performed according to standard surgical techniques routinely used in clinical practice.

The primary outcome of the study is laser efficiency, which will be evaluated using intraoperative laser system data,including grams of enucleated prostate tissue per joule (g/J). Preoperative prostate volume and intraoperative laser parameters are routinely recorded and will be used for analysis. No additional diagnostic procedures or treatments will be performed specifically for study purposes.

Secondary outcomes include changes in the International Prostate Symptom Score (IPSS) from preoperative assessment to postoperative follow-up and the presence of postoperative urinary incontinence. Safety assessment will be based on perioperative and postoperative adverse events recorded during routine clinical care.

The study will be conducted in accordance with ethical principles and applicable regulatory requirements, and patient confidentiality will be maintained throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with benign prostatic hyperplasia (BPH) and scheduled for anatomical prostate enucleation
* Presence of a prostate and clinical indication for surgical treatment
* Age between 50 and 80 years

Exclusion Criteria:

* History or suspicion of prostate cancer
* Previous prostate surgery
* Presence of neurogenic bladder or significant lower urinary tract dysfunction unrelated to BPH
* Active urinary tract infection at the time of surgery
* Severe comorbid conditions contraindicating surgery or anesthesia

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Individuals of any gender identity who have a prostate and meet the clinical eligibility criteria for prostate enucleation surgery are eligible to participate in this study.
Enrollment: 159 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Laser Enucleation Efficiency (g/J) | Intraoperative
  Laser enucleation efficiency will be evaluated by calculating the amount of enucleated prostate tissue in grams per joule of laser energy used (g/J), based on intraoperative laser system data and enucleated tissue weight recorded during surgery.

SECONDARY OUTCOMES:
Change in International Prostate Symptom Score (IPSS) | Baseline (preoperative) and 3 months postoperatively
  Change in the International Prostate Symptom Score (IPSS) from preoperative assessment to postoperative follow-up will be evaluated to assess functional outcomes after prostate enucleation.
Postoperative Urinary Incontinence | Up to 3 months postoperatively
  The presence of postoperative urinary incontinence will be assessed during routine postoperative follow-up visits.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Ilker Gokce, Prof., Principal Investigator — Ankara University
Locations (1):
- Ankara University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data that underlie the results reported in publications will be made available upon reasonable request.
Supporting Information: Study Protocol
Time Frame: Beginning 6 months after publication and ending 5 years after publication.
Access Criteria: Data will be shared with qualified researchers who provide a methodologically sound proposal. Requests should be directed to the corresponding investigator.